CLINICAL TRIAL: NCT02699151
Title: INvestigating SIGnificant Health TrendS in the Management of Superficial Vein Thrombosis (INSIGHTS-SVT)
Brief Title: INvestigating SIGnificant Health TrendS in the Management of Superficial Vein Thrombosis
Acronym: INSIGHTS-SVT
Status: Completed | Type: Observational
Sponsor: GWT-TUD GmbH (Other)
Responsible Party: Sponsor
Other Study IDs: INSIGHTS-SVT
Record Dates: First submitted 2016-01-21; First posted 2016-03-04 (Estimated); Last update posted 2023-09-14 (Actual); Status verified 2021-07

CONDITIONS: Superficial Vein Thrombosis
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: any drug — Any drug used for the treatment of SVT (e.g. heparin, low-molecular heparin, non-steroidal anti-inflammatory drug, fondaparinux, vitamin K antagonist)
Procedure: any procedure/surgery — Any procedure used for the treatment of SVT(e.g. sclerotherapy, endovenous thermotherapy, crossectomy, stripping, thrombectomy, phlebectomy)
Other: Any non-pharmacological treatment of SVT — Any non-pharmacological treatment of SVT (including watchful waiting)

SUMMARY:
Superficial vein thrombosis (SVT) and venous thromboembolism (VTE) are related entities. Only in the last years a series of observational studies mainly conducted in France could show that ´isolated SVT´ (without concomitant deep vein thrombosis and/or pulmonary embolism) is in fact not a benign and spontaneously healing disease but bears a potential for severe thromboembolic complications once not treated adequately. INSIGHTS-SVT study aims at collecting representative data on the current management and outcomes of SVT in Germany under real-life conditions. It will document the implementation of the recently issued national SVT guidelines issued by the Society for Angiology (DGA) and the Society for Phlebology (DGP).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed, acute, isolated SVT of the lower extremities
* written informed consent

Exclusion Criteria:

* SVT located at ≤ 3 cm of the saphenofemoral crossing (as such patients need to be treated for DVT)
* Subjects unlikely to comply with the requirements of the protocol (due to cognitive and/or language limitations)
* Patient(likely) not available for 1-year documentation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in hospital or ambulatory care
Sampling Method: Non-Probability Sample
Enrollment: 1210 (Actual)
Dates: Start 2016-04-14 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Efficacy: incidence of venous thromboembolism (VTE) events | 3 months
  VTE: composite of symptomatic pulmonary embolism (PE), symptomatic deep vein thrombosis (DVT), symptomatic recurrent superficial vein thrombosis (SVT), or symptomatic progression (extension) of SVT.
  This endpoint comprises symptomatic and asymptomatic VTE as reported by the treating physicians (usually diagnosed with compression ultrasonography or other appropriate methods).
  Events will be adjudicated.
Safety: incidence of major and clinically relevant bleeding events | 3 months
  Definition of bleeding events is based on American College of Chest Physicians Evidence-Based Clinical Practice Guidelines (major bleedings) and the "Comparison of Arixtra in lower limb superficial vein thrombosis with placebo" (CALISTO) study definition (other bleedings), respectively.
  Events will be adjudicated.

SECONDARY OUTCOMES:
Incidence of deep vein thrombosis (DVT) | 12 months
  Symptomatic and asymptomatic events as reported by the treating physician (usually diagnosed with compression ultrasonography or other appropriate methods).
  Events will be adjudicated.
Incidence of lung embolism (LE) | 12 months
  Symptomatic and asymptomatic events as reported by the treating physician. Events will be adjudicated.
Incidence of superficial vein thrombosis (SVT) | 12 months
  Symptomatic recurrent SVT: new occurrence of symptomatic SVT confirmed by compression ultrasonography or duplex-ultrasonography, in any other superficial vein.
  Symptomatic progression of initially diagnosed SVT: extension by at least 2 cm, confirmed compression ultrasonography or duplex ultrasonography, and > 3 cm away from the saphenofemoral crossing.
  Events will be adjudicated.
Death | 3 months and 12 months
New or recurrent cancer | 3 months and 12 months
VTE rates in the subgroup of patients who underwent surgical procedures for SVT | 3 months and 12 months
Predictors of VTE during follow-up | through study completion, up to 12 months
Diagnostic procedures for venous thromboembolism | through study completion, up to 12 months
  Utilisation rates of compression ultrasonography, duplex sonography, D-Dimer tests, computer tomography and other procedures typically used for the diagnosis of VTE.
Number of days in hospital due to VTE | through study completion, up to 12 months
Number of days spent in rehabilitation due to VTE | through study completion, up to 12 months
Numerical pain scale | through study completion, up to 12 months
  0-10 point scale
Health-related quality of life on Euroquol 5 Dimensions questionnaire | 3 months
  EQ-5D questionnaire
Health related quality of life on "VEnous Insufficiency Epidemiological and Economic Study" questionnaire | 3 months
  VEINES-QOL/Sym questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Rupert Bauersachs, MD, Principal Investigator — Gefäßzentrum, Klinikum Darmstadt; David Pittrow, MD, Study Director — GWT-TUD GmbH
Locations (1):
- Gefäßzentrum Darmstadt, Darmstadt, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bauersachs R, Gerlach HE, Heinken A, Hoffmann U, Langer F, Noppeney T, Pittrow D, Klotsche J, Rabe E; Collaborators. Rationale, design, and methodology of the observational INSIGHTS-SVT study on the current state of care and outcomes of patients with superficial vein thrombosis. J Vasc Surg Venous Lymphat Disord. 2017 Jul;5(4):553-560.e1. doi: 10.1016/j.jvsv.2017.03.013. PMID 28623995
- [Result] Bauersachs R, Gerlach HE, Heinken A, Hoffmann U, Langer F, Noppeney T, Pittrow D, Klotsche J, Rabe E. Management and Outcomes of Patients with Isolated Superficial Vein Thrombosis under Real Life Conditions (INSIGHTS-SVT). Eur J Vasc Endovasc Surg. 2021 Aug;62(2):241-249. doi: 10.1016/j.ejvs.2021.04.015. Epub 2021 Jun 29. PMID 34210599
- [Result] Rabe E, Hoffmann U, Schimke A, Heinken A, Langer F, Noppeney T, Pittrow D, Klotsche J, Gerlach HE, Bauersachs R; INSIGHTS-SVT Study Collaborators. Determinants of Late Venous Thromboembolic Events After Acute Isolated Superficial Vein Thrombosis in Daily Practice: 12 Month Results of the INSIGHTS-SVT Study. Eur J Vasc Endovasc Surg. 2023 Nov;66(5):697-704. doi: 10.1016/j.ejvs.2023.08.031. Epub 2023 Aug 12. PMID 37573936
- [Result] Langer F, Gerlach HE, Schimke A, Heinken A, Hoffmann U, Noppeney T, Pittrow D, Klotsche J, Rabe E, Bauersachs R; INSIGHTS-SVT study group. Clinical outcomes of cancer-associated isolated superficial vein thrombosis in daily practice. Thromb Res. 2022 Dec;220:145-152. doi: 10.1016/j.thromres.2022.10.022. Epub 2022 Nov 5. No abstract available. PMID 36370650